CLINICAL TRIAL: NCT01990300
Title: Long-term Use of Alogliptin/Pioglitazone Combination Tablets in Patients With Type 2 Diabetes Mellitus
Brief Title: Alogliptin/Pioglitazone (Liovel) Combination Tablets Survey on Long-term Use in Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 136-011; JapicCTI-132302 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin; Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alogliptin/Pioglitazone combination tablets: Alogliptin/Pioglitazone combination tablets, taken orally, once daily for up to 12 months. Participants received interventions as part of routine medical care.
  Interventions: Drug: Alogliptin/Pioglitazone

INTERVENTIONS:
Drug: Alogliptin/Pioglitazone — Alogliptin/Pioglitazone combination tablets
  Other Names: Liovel、SYR-322-4833

SUMMARY:
The purpose of this survey is to examine the safety and efficacy of long-term use of alogliptin/pioglitazone(Liovel) combination tablets in patients with type 2 diabetes mellitus determined as warranting combination therapy with alogliptin benzoate and pioglitazone hydrochloride

DETAILED DESCRIPTION:
This is a special drug use surveillance on long-term use of alogliptin/pioglitazone combination tablets. This study is designed to investigate the safety and efficacy of long-term use of alogliptin/pioglitazone combination tablet in patients with type 2 diabetes mellitus in the routine clinical setting.

Participants will be patients with type 2 diabetes mellitus. The planned sample size is 3000.

The usual adult dosage is 1 tablet (containing alogliptin/pioglitazone at either 25 mg/15 mg or 25 mg/30 mg) taken orally once daily before or after breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded:

  1. Patients with current cardiac failure or a past history of cardiac failure
  2. Patients with severe ketosis, diabetic coma or precoma, or type 1 diabetes mellitus
  3. Patients with serious hepatic dysfunction
  4. Patients with serious renal dysfunction
  5. Patients with severe infection, pre- or post-operative patients, or patients with serious traumatic injury
  6. Patients with a history of hypersensitivity to any ingredients of Alogliptin/Pioglitazone
  7. Pregnant or possibly pregnant women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus who have been examined at a medical institution
Sampling Method: Non-Probability Sample
Enrollment: 3281 (Actual)
Dates: Start 2011-11-28 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Someplace, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 445 investigative sites in Japan, from 28 November 2011 to 31 March 2015.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus were enrolled to receive Alogliptin/Pioglitazone 25 milligram (mg)/ 15 mg or 25 mg / 30 mg combination tablet orally, once daily for up to 12 months.
Groups:
- Alogliptin/Pioglitazone: Alogliptin/Pioglitazone 25 mg/ 15 mg or 25 mg/ 30 mg combination tablet, orally, once daily for up to 12 months in participants based upon the disease severity. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Alogliptin/Pioglitazone
Started | 3281
Completed | 3139
Not Completed | 142
Not completed — Case Report Forms Uncollected | 89
Not completed — Protocol Deviation | 53

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set; The safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Alogliptin/Pioglitazone
Number analyzed (Participants) | 3139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1188
  Male | 1951
Region of Enrollment [Number; unit: Participants]
  Japan | 3139
Duration of Type 2 Diabetes Mellitus [Mean (Standard Deviation); unit: Years] — Mean Duration between start of study and first time of diagnosis of type 2 diabetes mellitus was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 2689
    (all) | 7.56 (6.950)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  kilograms (kg)
    number analyzed (Participants) | 1982
    (all) | 68.87 (15.094)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/m^2
    number analyzed (Participants) | 1847
    (all) | 26.49 (4.592)
Waist Circumference (Male) [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in male participants.
  Participants
    number analyzed (Participants) | 1951
    <85 centimeter (cm) | 108
    ≥85cm | 317
    Unknown | 1526
Waist Circumference (Female) [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    number analyzed (Participants) | 1188
    <90cm | 146
    ≥90cm | 128
    Unknown | 914
Healthcare Category [Count of Participants; unit: Participants]
  Outpatient | 3113
  Inpatient | 26
Pregnancy Status (Not Pregnant) [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    number analyzed (Participants) | 1188
    (all) | 1188
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Presence of Medical Complications | 441
    Had Presence of Medical Complications | 2698
Diabetic Complications [Count of Participants; unit: Participants]
  Had No Presence of Diabetic Complications | 2621
  Had Presence of Diabetic Complications | 518
Concomitant Lifestyle-Related Disease [Count of Participants; unit: Participants]
  Had No Concomitant Lifestyle-Related Disease | 583
  Had Concomitant Lifestyle-Related Disease | 2556
Concomitant Hepatic Disorder [Count of Participants; unit: Participants]
  Had No Concomitant Hepatic Disorder | 2662
  Had Concomitant Hepatic Disorder | 477
Degree of Hepatic Dysfunction [Count of Participants; unit: Participants] — Severity was determined using aspartate aminotransferase (AST) or alanine transaminase (ALT) values at the start of treatment with alogliptin. For the assessment of severity, the following categories were used and higher grades of serum AST or ALT were adopted. Normal: <50 international units per liter (IU/L) Grade 1: >=50 to <100 IU/L Grade 2: >=100 to <500 IU/L Grade 3: >=500 IU/L
  Participants
    Normal | 1765
    Grade 1 | 216
    Grade 2 | 40
    Grade 3 | 1
    Unknown | 1117
Concomitant Renal Disorder [Count of Participants; unit: Participants]
  Had No Concomitant Renal Disorder | 2760
  Had Concomitant Renal Disorder | 379
Degree of Renal Dysfunction (eGFR) [Count of Participants; unit: Participants] — Estimated glomerular filtration rate (eGFR) was calculated using variables of gender, age at the start of treatment, and serum creatinine values, and severity was determined based on the following categories. If the serum creatinine value at the start of treatment was not listed, the severity was reported as "unknown." Normal: >=90 milliliter per min (mL/min)/1.73^2, Mild: >=60 mL/min/1.73^2 to <90 mL/min/1.73^2, Moderate: >=30 mL/min/1.73^2 to <60 mL/min/1.73^2, Severe: <30 mL/min/1.73^2 eGFR = 194 * Cr^-1.094 * (age)^-0.287 (* 0.739 if female) where Cr is creatinine value.
  Participants
    Normal | 462
    Mild | 1090
    Moderate | 411
    Severe | 21
    Unknown | 1155
Degree of Renal Dysfunction (Cr) [Count of Participants; unit: Participants] — Normal or Mild: =< 1.4 mg/dL (for male) or =< 1.2 mg/dL (for female), Moderate: >1.4 mg/dL to =< 2.4 mg/dL (for male) or >1.2 mg/dL to =< 2.0 mg/dL (for female), Severe: > 2.4 mg/dL (for male), > 2.0 mg/dL (for female). If the serum creatinine value (Cr) at the start of treatment was not listed, the severity was reported as "unknown."
  Participants
    Normal or Mild | 1933
    Moderate | 49
    Severe | 2
    Unknown | 1155
Concomitant Cardiac Disease [Count of Participants; unit: Participants]
  Had No Concomitant Cardiac Disease | 2828
  Had Concomitant Cardiac Disease | 311
Concomitant Heart Failure [Count of Participants; unit: Participants]
  Had No Concomitant Heart Failure | 3134
  Had Concomitant Heart Failure | 5
New York Heart Association (NYHA) Heart Failure Classification [Count of Participants; unit: Participants] — NYHA functional classification ranges from Class I (Participants with cardiac disease but without resulting limitations of physical activity), Class II (Cardiac disease resulting in slight limitation of physical activity), Class III (Cardiac disease resulting in marked limitation of physical activity), Class IV (Cardiac disease resulting in inability to carry on any physical activity without discomfort). Population: The baseline measure was analyzed only for participants who had complications of heart failure. Data of one participant was not collected throughout this study.
  Participants
    number analyzed (Participants) | 4
    Class I | 3
    Class II | 1
Concomitant Stroke-Related Disease [Count of Participants; unit: Participants]
  Had No Concomitant Stroke-Related Disease | 2979
  Had Concomitant Stroke-Related Disease | 160
Concomitant Allergic Condition [Count of Participants; unit: Participants]
  Had No Concomitant Allergic Condition | 2954
  Had Concomitant Allergic Condition | 185
Concomitant Malignant Tumor [Count of Participants; unit: Participants]
  Had No Concomitant Malignant Tumor | 3092
  Had Concomitant Malignant Tumor | 47
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had No Presence of Medical History | 2523
    Had Presence of Medical History | 347
    Unknown | 269
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had No Predisposition to Hypersensitivity | 2735
    Had Predisposition to Hypersensitivity | 119
    Unknown | 285
Drinking Habits [Count of Participants; unit: Participants]
  Current Drinker | 900
  Never Drank or Ex Drinker | 1538
  Unknown | 701
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 1260
  Current Smoker | 480
  Ex-Smoker | 557
  Unknown | 842
Haemoglobin A1c (HbA1c) [National Glycohemoglobin Standardization Program (NGSP)] [Mean (Standard Deviation); unit: Percent HbA1c] — Population: The number analyzed is the number of participants with data available for analysis.
  Percent HbA1c
    number analyzed (Participants) | 2909
    (all) | 7.63 (1.276)
Alogliptin Status [Count of Participants; unit: Participants]
  Had No Doses of Alogliptin | 2092
  Had Doses of Alogliptin | 1047
Pioglitazone Status [Count of Participants; unit: Participants]
  Had No Doses of Pioglitazone | 1402
  Had Doses of Pioglitazone | 1737

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Adverse Events
Time Frame: Up to 12 Months
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Alogliptin/Pioglitazone
Number analyzed (Participants) | 3139
Participants | 206

2. Primary Outcome: Changes From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: Reported data are changes in HbA1c from baseline at Month 1, 3, 6, 12 and final assessment (up to 12 months).
Time Frame: Baseline and Month 1, 3, 6, 12 and final assessment (up to 12 Months)
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. The number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Alogliptin/Pioglitazone
Number analyzed (Participants) | 2830
Percent HbA1c
  Change in HbA1c at Month 1: number analyzed (Participants) | 2094
  Change in HbA1c at Month 1 | -0.26 (0.651)
  Change in HbA1c at Month 3: number analyzed (Participants) | 2380
  Change in HbA1c at Month 3 | -0.58 (0.991)
  Change in HbA1c at Month 6: number analyzed (Participants) | 2404
  Change in HbA1c at Month 6 | -0.66 (1.081)
  Change in HbA1c at Month 12: number analyzed (Participants) | 2372
  Change in HbA1c at Month 12 | -0.66 (1.098)
  Change in HbA1c at Final Assessment | -0.65 (1.121)

3. Secondary Outcome: Changes From Baseline in Fasting Blood Glucose (FBG)
Description: Reported data are changes in fasting blood glucose level from baseline at Month 1, 3, 6, 12 and final assessment (up to 12 months).
Time Frame: Baseline and Month 1, 3, 6, 12 and final assessment (up to 12 Months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin/Pioglitazone
Number analyzed (Participants) | 1554
mg/dL
  Change in FBG at Month 1: number analyzed (Participants) | 1052
  Change in FBG at Month 1 | -14.7 (49.34)
  Change in FBG at Month 3: number analyzed (Participants) | 1195
  Change in FBG at Month 3 | -18.7 (50.24)
  Change in FBG at Month 6: number analyzed (Participants) | 1243
  Change in FBG at Month 6 | -18.4 (50.51)
  Change in FBG at Month 12: number analyzed (Participants) | 1239
  Change in FBG at Month 12 | -19.6 (50.93)
  Change in FBG at Final Assessment | -19.8 (53.31)

ADVERSE EVENTS:
Time Frame: Up to Month 12
Description: At each visit the investigator had to document any occurrence of adverse drug reactions (ADRs). Any events reported by the participant or observed by the investigator were recorded, irrespective of the relation to study treatment. Only ADRs were collected in this study. Participants may be represented in more than 1 category.
Arm/Group | Alogliptin/Pioglitazone
Serious Adverse Events (participants affected / at risk) | 4/3139
Other Adverse Events (participants affected / at risk) | 56/3139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin/Pioglitazone (N=3139)
Pneumonia (Infections and infestations) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin/Pioglitazone (N=3139)
Rash (Skin and subcutaneous tissue disorders) | 5
Oedema (General disorders) | 32
Oedema peripheral (General disorders) | 8
Weight increased (Investigations) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.